CLINICAL TRIAL: NCT00407719
Title: An Open-Label, Pilot Study of Bevacizumab in Subjects With Choroidal Neovascularization Secondary to Diseases Other Than Age-Related Macular Degeneration
Brief Title: Bevicizumab (Avastin) Infusion for Choroidal Neovascularization (CNV) Not Associated With Age-Related Macular Degeneration (AMD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Quan Dong Nguyen, MD, MSc, Johns Hopkins University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FVF 3687; 05-05-16-06
Record Dates: First submitted 2006-12-01; First posted 2006-12-05 (Estimated); Last update posted 2009-02-03 (Estimated); Status verified 2009-01

CONDITIONS: Choroidal Neovascularization; Degenerative Myopia; Pathological Myopia
Keywords: Choroidal Neovascularization
MeSH Terms: conditions — Choroidal Neovascularization; Myopia, Degenerative | interventions — Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab

SUMMARY:
The purpose of this study is to see if the drug bevacizumab is safe and effective to use for people with choroidal neovascularization (CNV). CNV is an eye condition where abnormal blood vessels grow in the part of the eye responsible for central (straight ahead) vision. The drug is produced using recombinant DNA technology and has been approved by the FDA for use in colon cancer. Although not yet approved for people with CNV, the FDA has given permission to use this drug in this study.

DETAILED DESCRIPTION:
Bevacizumab is a recombinant humanized monoclonal antibody against VEGF. It has been approved by the FDA for the treatment of metastatic colon cancer 18. We hypothesize that VEGF also plays a role in the development of CNV in pathologic myopia. Therefore, employing a mode of therapy that would decrease the risks posed to eyes with attenuated sclera, we have treated, through special approval by the Pharmacy and Therapeutic Committee of the Johns Hopkins University School of Medicine, two patients with persistent myopic CNV with intravenous bevacizumab 19. Despite multiple treatments with PDT, the CNV remained active and vision continued to decline in these two index patients. After four infusions of bevacizumab, the CNV became inactive. Six months after the last infusion in each patient, the CNV showed no evidence of activity or leakage on fluorescein angiography. Vision also improved in the diseased eyes of both patients. The two patients tolerated the infusions well, with no adverse events detected. In particular, blood pressure remained stable and no proteinuria was noted on serial analyses of 24-hour urine collections. The Bascom Palmer Eye Institute at the University of Miami has also recently reported favorable outcomes of bevacizumab administered in repeated doses to 14 patients (age > 65 years) with CNV secondary to AMD that has been refractory to other therapies.

We propose a non-randomized, open-label pilot study to evaluate the effect of bevacizumab in patients with CNV due to any cause other than AMD. This design will allow us to closely monitor safety and tolerability of bevacizumab while we evaluate 3 bioactivity outcomes. Based upon dramatic responses in two patients with CNV due to myopic degeneration, we hypothesize that treatment with bevacizumab may have major advantages over current standard of care.

ELIGIBILITY:
Abbreviated: Contact Coordinator or Principal investigator for expanded criteria.

Inclusion Criteria:) Subfoveal CNV in study eye due to cause other than AMD. Best corrected visual acuity of 20/30 or less in study eye. Evidence of retinal thickening or subretinal fluid by OCT in study eye. Must be fluorescein leakage due to CNV in the study eye. If the CNV is a complication of another disease (i.e. uveitis), the disease must be under stabilization for at least 3 months prior to enrollment.

(ECG)at least 28 days prior to entry into the study must show no evidence of current or prior myocardial ischemia, infarction, or significant arrhythmia.

Adequate bone marrow function:

Absolute granulocyte count (neutrophils and bands) > 1500 cells/mm3;

1. Platelet count > 100,000 cells/mm3;
2. 9.0 g/dL; 9) PT/PTT within the institution upper limit of Hemoglobin, normal (ULN) or INR <1.1. 10) Adequate renal function: serum creatinine ≤ 2.0 mg/dL. 11)Patients of child bearing potential must abstain from sexual intercourse or use effective birth control. Negative serum pregnancy test result confirmation prior to treatment.

Patients must be able to return for all study visits within required visit windows.

Patients must provide written informed consent

- Exclusion Criteria:

1. Previous subfoveal thermal laser therapy.
2. Significant scarring or atrophy in the fovea that indicates substantial irreversible vision loss.
3. Significant media opacities, including cataract, which can interfere with visual acuity, assessment of toxicity, or fundus photography.
4. Any intraocular surgery in the study eye within 12 weeks of entry.
5. If the CNV in the study eye has been treated with photodynamic therapy (PDT), the treatment must be at least 12 weeks prior to study entry, unless it is judged by the investigator that the ocular disease has deteriorated within the 12-week period
6. Any treatment for CNV in the study eye with anti-vascular endothelial growth factor (anti-VEGF) therapy, intraocularly or intravenously, must be at least 6 weeks prior to study entry, unless it is judged that the ocular disease has deteriorated within the 6-week period
7. Uncontrolled hypertension defined as blood pressure consistently (at 3 or more consecutive visits) greater than 150/100 irrespective or medication.
8. Any history, physical signs, or EKG findings suggesting significant heart disease.
9. History of thromboembolism or stroke.
10. History, physical signs, or laboratory of bleeding diathesis or coagulopathy. Any history (within 3 years) of significant gastrointestinal, oral (gum), or nasal bleeding..
11. History or physical signs of peripheral vascular disease.
12. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to entry.
13. Anticipation of need for major surgical procedure during the course of the study.
14. Minor surgical procedures, fine needle aspirations or core biopsies within 7 days prior to entry.
15. Women who are pregnant (positive pregnancy test) or breastfeeding.
16. Protein concentration in a 24-hour urine specimen more than 1.3 x ULN.
17. History of abdominal fistula, gastrointestinal perforation, or intra- abdominal abscess within 6 months prior to entry.
18. Serious, non-healing wound, ulcer, or bone fracture.
19. Lung carcinoma of squamous cell histology or any histology in close proximity to a major vessel, cavitation, or history of hemoptysis.
20. Inability to comply with study and/or follow-up procedures.
21. Any patient who is on standard anticoagulant therapy [INR targeted at 2.0 to 3.0] or treatment for deep vein thrombosis, or grade 3 or 4 venous thrombosis (Table 1), is not eligible to enroll in the study. Patients who are on stable, low-dose heparin or warfarin therapy may be eligible for the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10
Dates: Start 2005-06; Primary Completion 2007-04 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Visual acuity: In this pilot study, the sample size is not powered for clinical response. However, preliminary data on visual acuity will aid in the design of future randomized control trial. | each visit for study duration up to 24 mos

SECONDARY OUTCOMES:
Retinal thickness assessed by OCT | each visit
CNV leakage assessed by Digital Fluorescein Angiography | per protocol

CONTACTS AND LOCATIONS:
Overall Officials: Quan D Nguyen, MD, MSc, Principal Investigator — Johns Hopkins University

REFERENCES:
- [Derived] Nguyen QD, Shah SM, Hafiz G, Do DV, Haller JA, Pili R, Zimmer-Galler IE, Janjua K, Symons RC, Campochiaro PA. Intravenous bevacizumab causes regression of choroidal neovascularization secondary to diseases other than age-related macular degeneration. Am J Ophthalmol. 2008 Feb;145(2):257-266. doi: 10.1016/j.ajo.2007.09.025. Epub 2007 Dec 11. PMID 18054887